CLINICAL TRIAL: NCT04343950
Title: Implementation of Text Messaging (SMS) as an Improvement Tool in Population-based Cancer Screening Programs
Brief Title: SMS Messaging as a Tool to Improve Cancer Screening Programs
Acronym: M-TICS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Català d'Oncologia (Other)
Collaborators: University of Dundee (Other); University of Barcelona (Other); University Rovira i Virgili (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: ICO_UCC_202001; PI19/00226 (Other Grant/Funding Number: The National Institute of Health Carlos III (ISCIII))
Record Dates: First submitted 2020-04-09; First posted 2020-04-14 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Mass Screening; Colorectal Cancer; Breast Cancer
Keywords: Uptake; Participation; Cost-effectiveness; Breast cancer screening; Colorectal cancer screening; Text-message; Mobile-health
MeSH Terms: conditions — Colorectal Neoplasms; Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Intervention 1: SMS reminders for colorectal cancer screening compared to reminder letters.
  Intervention 2: SMS reminders to return the fecal occult blood test at the pharmacy compared to no intervention.
  Intervention 3: Invitation by SMS for women with a prior participation in the breast cancer screening program compared to invitation letter.
Masking Description: Invited individuals to the cancer screening programs will not be aware of the different arms of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Intervention 1: SMS reminders in colorectal cancer screening (Experimental): SMS reminders will be sent to individuals who received an invitation letter from Colorectal Cancer Screening Program and haven't participated within 6 weeks.
  Interventions: Behavioral: SMS reminders to enhance colorectal cancer screening
- Usual Care 1: Reminder letter in colorectal cancer screening (Active Comparator): Reminder letters will be sent to individuals who received an invitation letter from the Colorectal Cancer Screening Program and haven't participated within 6 weeks.
  Interventions: Behavioral: SMS reminders to enhance colorectal cancer screening
- Intervention 2: SMS reminders to return the screening test (Experimental): SMS reminders will be sent to individuals who picked the fecal immunochemical test at the pharmacy and haven't returned it within 14 days.
  Interventions: Behavioral: SMS reminders to return the fecal immunochemical test at the pharmacy in CRC screening:
- Usual Care 2: No intervention (Active Comparator): No reminders will be sent.
  Interventions: Behavioral: SMS reminders to return the fecal immunochemical test at the pharmacy in CRC screening:
- Intervention 3: SMS invitation among prior participants (Experimental): Invitation by SMS will be sent to women who previously participated in the Breast Cancer Screening Program.
  Interventions: Behavioral: Invitation by SMS to previous participants in breast cancer screening:
- Usual Care 3: Invitation letter (Active Comparator): Letter invitations will be sent.
  Interventions: Behavioral: Invitation by SMS to previous participants in breast cancer screening:

INTERVENTIONS:
Behavioral: SMS reminders to enhance colorectal cancer screening — Individual randomization will be used. Individuals assigned to the experimental arm with a wrong phone number will get a reminder letter (protocol analysis).
  Other Names: Intervention 1
  Arms: Intervention 1: SMS reminders in colorectal cancer screening; Usual Care 1: Reminder letter in colorectal cancer screening
Behavioral: SMS reminders to return the fecal immunochemical test at the pharmacy in CRC screening: — Individual randomization will be used. Individuals with a wrong phone number assigned to the experimental arm will not get any reminder (protocol analysis).
  Other Names: Intervention 2
  Arms: Intervention 2: SMS reminders to return the screening test; Usual Care 2: No intervention
Behavioral: Invitation by SMS to previous participants in breast cancer screening: — Individual randomization. Women assigned to the experimental arm and with a wrong phone number will get an invitation letter (protocol analysis).
  Other Names: Intervention 3
  Arms: Intervention 3: SMS invitation among prior participants; Usual Care 3: Invitation letter

SUMMARY:
The aim of this project is to assess the impact on health and economics of the implementation of text messaging (SMS) in cancer screening programs. Three interventions with SMS will be evaluated through community trials. In the colorectal cancer screening program the following interventions will be tested: a) Participation reminder: six weeks after sending the invitation letter of the colorectal cancer program if there has not been a response, a reminder SMS will be sent in front of the usual method by letter; b) Reminder to return the fecal occult blood test: SMS reminder of test delivery versus no intervention. This reminder will be sent to the individuals who have gone to the pharmacy to pick up a fecal occult blood test and they have not returned it after 14 days. The impact on participation will be analyzed and, if applicable, the proportion of advanced neoplasms will be calculated by increase in participation. In the breast cancer screening program, the invitation by SMS versus the usual invitation by letter will be studied in women who had participated in the previous screening round. The impact on participation will be analyzed. A cost-effectiveness analysis of the three interventions will be carried out. The incremental cost ratio of the interventions between cost variation and effectiveness variation will be calculated.

DETAILED DESCRIPTION:
Main Hypothesis:

The implementation of SMS in population-based cancer screening programs will improve participation, especially in colorectal cancer screening, will allow a better resource management and reduce costs in both programs.

Specific Hypothesis:

Sending the reminder SMS will have an impact on participation greater than that obtained with the standard reminder (letter) in the colorectal cancer screening program.

The effect of the colorectal cancer screening reminder SMS will be greater among the individuals who have been invited for the first time and not previous participants.

Participation after receiving the invitation by SMS in breast cancer screening will be equal to or better than the letter invitation.

The alternative that includes sending SMS will be cost-effective in relation to the current alternative that you use postal shipping.

ELIGIBILITY:
Inclusion Criteria:

* Eligible individuals for colorectal cancer screening (intervention 1 and 2)
* Eligible women for breast cancer screening (intervention 3)
* Registered at the HealthCare Database (RCA)

Exclusion Criteria:

* Individuals without a mobile phone number registered at the RCA
* Opt out from breast cancer screening and/or colorectal cancer screening

Ages: 50 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Intervention 1 and 2: both sexes. Intervention 3: only women.
Enrollment: 44601 (Actual)
Dates: Start 2021-06-05 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Intervention 1: Participation in colorectal cancer screening program | 18 weeks
  Participation (no/yes) will be gathered prospectively 18 weeks after sending the screening invitation letter (week 0).
Intervention 2: Participation in colorectal cancer screening program among individuals who pick the test at the pharmacy | 18 weeks
  Participation (no/yes) among those individuals who pick the screening test for colorectal cancer at the pharmacy 18 weeks after sending the screening invitation letter (week 0).
Intervention 3: Participation in breast cancer screening program | 8 weeks
  Participation (no/yes) will be gathered prospectively 8 weeks after sending the screening invitation letter (week 0).

SECONDARY OUTCOMES:
Incremental cost ratio | 18 weeks
  A cost-effectiveness analysis of the three interventions will be carried out. The incremental cost ratio of the interventions between cost variation and effectiveness variation will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Montse Garcia, PhD, Principal Investigator — Institut Català d'Oncologia
Locations (1):
- Institut Català d'Oncologia, L'Hospitalet de Llobregat, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vives N, Binefa G, Travier N, Farre A, Panera JA, Casas B, Vidal C, Ibanez-Sanz G, Garcia M; M-TICS research group. Text Messaging Versus Postal Reminders to Improve Participation in a Colorectal Cancer Screening Program: Randomized Controlled Trial. JMIR Mhealth Uhealth. 2025 Jan 1;13:e64243. doi: 10.2196/64243. PMID 39742454
- [Background] Vives N, Vidal C, de Guzman EN, Farre A, Panera JA, Binefa G, Garcia M; M-TICS research group. The use of text messages as an alternative invitation method for breast cancer screening: A randomized controlled trial (M-TICS study). PLoS One. 2024 Aug 29;19(8):e0306720. doi: 10.1371/journal.pone.0306720. eCollection 2024. PMID 39208325
- [Background] Vives N, Travier N, Farre A, Binefa G, Vidal C, Perez Lacasta MJ, Ibanez-Sanz G, Nino de Guzman EP, Panera JA, Garcia M; M-TICS Research Group. Effectiveness and Acceptability of Targeted Text Message Reminders in Colorectal Cancer Screening: Randomized Controlled Trial (M-TICS Study). JMIR Public Health Surveill. 2024 Jul 31;10:e57959. doi: 10.2196/57959. PMID 39083331
- [Background] Vives N, Farre A, Ibanez-Sanz G, Vidal C, Binefa G, Mila N, Perez-Lacasta MJ, Travier N, Benito L, Espinas JA, Bagaria G, Garcia M. Text messaging as a tool to improve cancer screening programs (M-TICS Study): A randomized controlled trial protocol. PLoS One. 2021 Jan 22;16(1):e0245806. doi: 10.1371/journal.pone.0245806. eCollection 2021. PMID 33481914